CLINICAL TRIAL: NCT06385977
Title: Risk Factors for Chronic Prostatitis/Chronic Pelvic Pain Syndrome Patients in Northwest China
Brief Title: Risk Factors for Chronic Prostatitis Patients in Northwest China
Status: Recruiting | Type: Observational
Sponsor: Shaanxi Provincial People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: ShaanxiPPH
Record Dates: First submitted 2024-04-24; First posted 2024-04-26 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Chronic Prostatitis With Chronic Pelvic Pain Syndrome
MeSH Terms: conditions — Prostatitis | interventions — Dosage Forms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- case group: participates diagnosed with Chronic prostatitis/chronic pelvic pain syndrome
  Interventions: Behavioral: lifestyle; Behavioral: sexual habits; Drug: medication
- control group: participates without Chronic prostatitis/chronic pelvic pain syndrome
  Interventions: Behavioral: lifestyle; Behavioral: sexual habits; Drug: medication

INTERVENTIONS:
Behavioral: lifestyle — Life habits and personal preferences
Behavioral: sexual habits — Sexual experience and activities
Drug: medication — use of medication

SUMMARY:
The goal of this observational study is to learn about the risk factors of lifestyle, medication and sexual habits in adult chronic prostatitis / chronic pelvic pain syndrome patients. The main questions it aims to answer are:

* Is lifestyle, medication, and sexual habits related to chronic prostatitis / chronic pelvic pain syndrome
* Is there any medication available to protect men from chronic prostatitis / chronic pelvic pain syndrome.

Participants will:

* Independently receive a survey questionnaire on lifestyle, medication, and sexual habits.
* Symptomatic individuals will undergo additional prostate fluid examination for diagnosis.

Researchers will compare healthy adult males to see if there are differences on lifestyle, medication and sexual habits between the two groups.

DETAILED DESCRIPTION:
All participants were asked to fill out a questionnaire which was modified based on Zhang Ran's research. The questionnaire contained the following parts: patient's general situation, dietary habits, disease status, medication, lifestyle, sexual habits and NIH-CPSI index (National Institutes of Health Chronic Prostatitis Symptom Index). Furthermore, the patients underwent digital rectal examination, expressed prostatic secretion microscopy and microbial culture, urinalysis, urine microbial culture and transrectal ultrasonography.

ELIGIBILITY:
Inclusion Criteria:

* Discomfort or pain in the pelvic region or perineum;
* Symptoms lasting for at least 3 months;
* NIH-CPSI pain score of ≥ 4;
* Controls are volunteers who do not present any prostatitis-related symptoms.

Exclusion Criteria:

* Prostate cancer;
* Benign prostatic hyperplasia with a post-void residual urine volume of >50 ml;
* Acute urinary tract infection.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients are from Urology Clinic, while all the controls are recruited from the physical examination center of our hospital.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2016-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Odds Ratio | baseline
  The ratio of exposed to unexposed individuals in the case group divided by the ratio of exposed to unexposed individuals in the control group

CONTACTS AND LOCATIONS:
Overall Officials: Chun Du, Professor, Study Director — Shaanxi Provincial People's Hospital
Locations (1):
- Shaanxi Provincial People's Hospital, Xi'an, Shaanxi, China